CLINICAL TRIAL: NCT02564523
Title: A Randomized, Observer-blind, Placebo-controlled, Phase 2 Study to Evaluate the Safety, Tolerability and Immunogenicity of Different Prime-boost Regimens of the Candidate Prophylactic Vaccines for Ebola Ad26.ZEBOV and MVA-BN-Filo in Healthy Adults, Including Elderly Subjects, HIV-infected Subjects, and Healthy Children in Two Age Strata in Africa
Brief Title: Safety, Tolerability and Immunogenicity Study of 3 Prime-boost Regimens for Ebola Vaccines Ad26.ZEBOV/MVA-BN-Filo in Healthy Adults, Children and Human Immunodeficiency Virus Positive (HIV+) Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: EBOVAC2 Consortium (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Muraz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR107249; VAC52150EBL2002 (Other: Janssen Vaccines & Prevention B.V.); 2019-000690-22 (EudraCT Number)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Hemorrhagic Fever, Ebola
Keywords: Healthy; Vaccine; Ebola viruses; Ebola virus disease (EVD); Filoviruses; Hemorrhagic fever; Monovalent vaccine; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic (MVA-BN) Filo-vector; Safety; Immunogenicity; Inserm, Centre Muraz
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive Ad26.ZEBOV, MVA-BN-Filo (Day 1/Day 29) or placebo (Day 1/Day 29) followed by a subset of participants who received Ad26.ZEBOV and MVA-BN-Filo (at selected sites) will receive Ad26.ZEBOV as third vaccination and who received placebo will receive placebo as third vaccination (at least 1 year post prime vaccination).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo
- Group 2 (Experimental): Participants will receive Ad26.ZEBOV, MVA-BN-Filo (Day 1/Day 57) or placebo (Day 1/Day 57) followed by a subset of participants who received Ad26.ZEBOV and MVA-BN-Filo (at selected sites) will receive Ad26.ZEBOV as third vaccination and who received placebo will receive placebo as third vaccination (at least 1 year post prime vaccination).
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo
- Group 3 (Experimental): Participants will receive Ad26.ZEBOV, MVA-BN-Filo (Day 1/Day 85) or placebo (Day 1/Day 85)
  Interventions: Biological: Ad26.ZEBOV; Biological: MVA-BN-Filo; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV — One 0.5 mL intramuscular (IM) injection of (5x10*10 viral particles)
Biological: MVA-BN-Filo — One 0.5 mL IM injection of (1x10*8 infectious units)
Biological: Placebo — One 0.5 mL IM injection of 0.9% saline

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of three heterologous prime-boost regimens for Ebola vaccines Ad26.ZEBOV and MVA-BN-Filo. The study will include healthy adults and elderly participants, HIV infected participants and healthy children in 2 age strata.

DETAILED DESCRIPTION:
This is a randomized, observer-blind, placebo-controlled, parallel-group, multicenter, Phase 2 study evaluating the safety, tolerability and immunogenicity of 3 heterologous prime-boost regimens using Ad26.ZEBOV as prime and MVA-BN-Filo as boost vaccination, administered at 28-, 56- and 84-day (Group 1, 2 and 3 as above) intervals, in healthy adults and elderly participants. A 28- and 56-day (Groups 1 and 2, as above) schedule will be evaluated in HIV-infected participants and in healthy children in 2 age strata. The study consists of a screening phase of up to 8 weeks, a vaccination phase in which participants will be vaccinated at baseline (Day 1) followed by a boost vaccination on Day 29, 57 or 85, a post-vaccination phase and long-term follow-up phase until Day 365. Participants in Cohort 1 substudy (Group 1 and 2) who received Ad26.ZEBOV and MVA-BN-Filo (at selected sites) will receive Ad26.ZEBOV as third vaccination and who received placebo will receive placebo as third vaccination (at least 1 year post prime vaccination). All participants within a cohort will be followed in a blinded manner by the site until the last subject in that cohort has completed the study. This study will be conducted in Africa and the enrollment will take place sequentially in three cohorts: the first cohort will consist of healthy participants (18 - 70 years); the second cohort (2a) will include HIV-infected participants (18 to 50 years) and healthy children 12 to 17 years (cohort 2b); the third cohort will include children aged 4 to 11 years inclusive will be enrolled. Within each cohort, participants will be randomized in a 5:1 ratio to receive active vaccine versus placebo. Safety evaluations will include assessments of adverse events, an electrocardiogram (ECG) for adult participants at screening, physical examination, vital signs (blood pressure, pulse/heart rate, body temperature), clinical laboratory and pregnancy testing. An independent data monitoring committee (IDMC) will be established to monitor data on a regular basis to ensure the continuing safety of the participants enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

Criteria for healthy adults and elderly participants:

* Participant must be healthy in the investigator's clinical judgment on the basis of clinical laboratory tests, medical history, ECG, physical examination and vital signs performed at screening. Participants with hemoglobin values outside the local laboratory reference ranges may be included if the hemoglobin is above the age/gender specific limits
* Female participants of childbearing potential must use adequate birth control measures, must have a negative pregnancy test at screening and immediately prior to each study vaccination
* A man who is sexually active with a woman of childbearing potential must be willing to use condoms for sexual intercourse beginning prior to enrollment, unless a vasectomy was performed more than 1 year prior to screening
* Participant must pass the test of understanding (TOU)
* Participant must be available and willing to participate for the duration of the study visits and follow-up, provide verifiable identification, and have a means to be contacted Additional Inclusion Criteria HIV-infected Participants
* Participant must be between 18 to 50 years of age and must have a documented HIV-infection for at least 6 months prior to screening
* Participant must be on a stable 3 drug regimen of Highly Active Antiretroviral Therapy for at least 4 weeks prior to screening and having a CD4 positive cell count of >350 cells/microliter. Also participant must be in an otherwise reasonable good medical condition Additional Inclusion Criteria Children Participants
* Parent/legal guardian must pass the TOU before signing the inform consent form. Informed assent must be obtained from adolescents and older children, depending on local regulations and practice
* Pediatric participant's age on the day of randomization must be within one of the 2 age strata: 12-17 years or 4-11 years (all ages inclusive)
* Pediatric participants must have received all routine immunizations appropriate for his or her age as reported by the parent(s)/legal guardian, according to local routine vaccination schedules

Exclusion criteria:

* Diagnosed with Ebola virus disease or previously exposed to Ebola virus including travel to epidemic Ebola areas less than 1 month prior to screening
* Having received any candidate Ebola vaccine or any experimental candidate Ad26- or MVA-based vaccine in the past
* Having HIV type 1 or type 2 infection (for healthy adults/elderly/children)
* Pediatric participants with weight-per-height below 10th percentile according to the Centers for Disease Control and Prevention (CDC) growth charts (4- to 11-year-olds)
* A woman who is pregnant, breast-feeding or planning to become pregnant while enrolled in the study or within at least 3 months after the prime vaccination or up to 1 month after the boost vaccination (whichever takes longer) or within at least 3 months after the third vaccination
* For HIV+ adults, no AIDS-defining illnesses

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1075 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (7):
- Burkina Faso (2):
  - BoboDioulasso
  - Ouagadougou
- Côte d’Ivoire (2):
  - Abidjan
  - Toupah/Ousrou
- Nairobi, Kenya
- Uganda (2):
  - Entebbe
  - Kampala

REFERENCES:
- [Derived] Barry H, Lhomme E, Surenaud M, Nouctara M, Robinson C, Bockstal V, Valea I, Somda S, Tinto H, Meda N, Greenwood B, Thiebaut R, Lacabaratz C. Helminth exposure and immune response to the two-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccine regimen. PLoS Negl Trop Dis. 2024 Apr 11;18(4):e0011500. doi: 10.1371/journal.pntd.0011500. eCollection 2024 Apr. PMID 38603720
- [Derived] Anywaine Z, Barry H, Anzala O, Mutua G, Sirima SB, Eholie S, Kibuuka H, Betard C, Richert L, Lacabaratz C, McElrath MJ, De Rosa SC, Cohen KW, Shukarev G, Katwere M, Robinson C, Gaddah A, Heerwegh D, Bockstal V, Luhn K, Leyssen M, Thiebaut R, Douoguih M; EBL2002 Study group. Safety and immunogenicity of 2-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccination in children and adolescents in Africa: A randomised, placebo-controlled, multicentre Phase II clinical trial. PLoS Med. 2022 Jan 11;19(1):e1003865. doi: 10.1371/journal.pmed.1003865. eCollection 2022 Jan. PMID 35015777
- [Derived] Barry H, Mutua G, Kibuuka H, Anywaine Z, Sirima SB, Meda N, Anzala O, Eholie S, Betard C, Richert L, Lacabaratz C, McElrath MJ, De Rosa S, Cohen KW, Shukarev G, Robinson C, Gaddah A, Heerwegh D, Bockstal V, Luhn K, Leyssen M, Douoguih M, Thiebaut R; EBL2002 Study group. Safety and immunogenicity of 2-dose heterologous Ad26.ZEBOV, MVA-BN-Filo Ebola vaccination in healthy and HIV-infected adults: A randomised, placebo-controlled Phase II clinical trial in Africa. PLoS Med. 2021 Oct 29;18(10):e1003813. doi: 10.1371/journal.pmed.1003813. eCollection 2021 Oct. PMID 34714820

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1075 participants were enrolled. Among 1075 participants, 1 participant was enrolled twice and 1 participant was enrolled erroneously, but did not receive any study vaccination.
Groups:
- Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval: Participants (healthy adults and elderly) received intramuscular (IM) injection of Ad26.ZEBOV 5*10^10 viral particles (vp) on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 infectious units (Inf.U) on Day 29. Subset of participants who earlier received Ad26.ZEBOV and MVA-BN-Filo (at selected sites), afterwards received IM injection of Ad26.ZEBOV 5*10^10 vp as a booster dose at 1 year post dose 1 (Day 365).
- Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval: Participants (healthy adults and elderly) received IM injection of Placebo 0.9 percent (%) saline on Day 1 followed by IM injection of placebo 0.9 % saline on Day 29. Subset of participants who earlier received placebo(at selected sites), afterwards received IM injection of placebo 0.9 % saline as a booster dose at 1 year post dose 1 (Day 365).
- Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval: Participants (healthy adults and elderly) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo Inf.U on Day 57. Subset of participants who earlier received Ad26.ZEBOV and MVA-BN-Filo (at selected sites), afterwards received IM injection of Ad26.ZEBOV 5*10^10 vp as a booster dose at 1 year post dose 1 (Day 365).
- Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval: Participants (healthy adults and elderly) received placebo 0.9% saline on Day 1 followed by IM injection of placebo 0.9% saline on Day 57. Subset of participants who earlier received Placebo (at selected sites), afterwards received IM injection of Placebo 0.9 % saline as a booster dose at 1 year post dose 1 (Day 365).
- Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval: Participants (healthy adults and elderly) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 85.
- Cohort 1: Placebo, Placebo, 84-Day Interval: Participants (healthy adults and elderly) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 85.
- Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval: Participants (human immunodeficiency virus [HIV]-infected adults) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 29.
- Cohort 2a: Placebo, Placebo, 28-Day Interval: Participants (HIV-infected adults) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 29.
- Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval: Participants (HIV-infected adults) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 57.
- Cohort 2a: Placebo, Placebo, 56-Day Interval: Participants (HIV-infected adults) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 57.
- Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval: Participants (Healthy Adolescents [12-17 years]) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 29.
- Cohort 2b: Placebo, Placebo, 28-Day Interval: Participants (Healthy Adolescents [12-17 years]) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 29.
- Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval: Participants ((Healthy Adolescents [12-17 years]) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 57.
- Cohort 2b: Placebo, Placebo, 56-Day Interval: Participants (Healthy Adolescents [12-17 years]) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 57.
- Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval: Participants (Healthy Children [4-11 years]) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 29.
- Cohort 3: Placebo, Placebo, 28-Day Interval: Participants (Healthy Children [4-11 years]) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 29.
- Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval: Participants (Healthy Children [4-11 years]) received IM injection of Ad26.ZEBOV 5*10^10 vp on Day 1 followed by IM injection of MVA-BN-filo 1*10^8 Inf.U on Day 57.
- Cohort 3: Placebo, Placebo, 56-Day Interval: Participants (Healthy Children [4-11 years]) received IM injection of Placebo 0.9 % saline on Day 1 followed by IM injection of Placebo 0.9 % saline on Day 57.
Period: Overall Study
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Started | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants Who Received Booster Dose at 1 Year Post Dose 1 (on Day 365) | 34 | 8 | 39 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 215 | 40 | 214 | 43 | 106 | 22 | 56 | 12 | 59 | 12 | 52 | 10 | 53 | 10 | 54 | 12 | 54 | 11
Not Completed | 10 | 3 | 10 | 1 | 4 | 0 | 3 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval | Total
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12 | 1073
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (12.41) | 32 (10.43) | 33.3 (11.52) | 33.3 (11.57) | 31.4 (11.53) | 33.7 (12.31) | 38.8 (6.61) | 34.3 (7.66) | 39 (6.69) | 42.1 (4.96) | 14.4 (1.76) | 14.5 (1.86) | 14.1 (1.56) | 14.2 (1.81) | 7.6 (2.06) | 7.1 (2.07) | 7.8 (2.23) | 7.3 (2.09) | 28.3 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 15 | 71 | 16 | 27 | 8 | 39 | 8 | 42 | 10 | 25 | 5 | 26 | 4 | 27 | 5 | 28 | 5 | 434
  Male | 152 | 28 | 153 | 28 | 83 | 14 | 20 | 4 | 17 | 2 | 30 | 6 | 29 | 6 | 27 | 7 | 26 | 7 | 639
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 9
  Not Hispanic or Latino | 222 | 42 | 222 | 43 | 110 | 21 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 53 | 12 | 53 | 12 | 1063
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 223 | 42 | 224 | 43 | 109 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12 | 1068
  White | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  BURKINA FASO | 76 | 16 | 73 | 16 | 30 | 1 | 16 | 4 | 14 | 2 | 26 | 5 | 29 | 4 | 25 | 5 | 23 | 4 | 369
  COTE D'IVOIRE | 38 | 9 | 44 | 6 | 22 | 7 | 8 | 1 | 11 | 2 | 0 | 0 | 0 | 0 | 12 | 3 | 12 | 3 | 178
  KENYA | 28 | 3 | 27 | 5 | 16 | 4 | 14 | 4 | 12 | 3 | 12 | 3 | 13 | 2 | 5 | 1 | 5 | 1 | 158
  UGANDA | 83 | 15 | 80 | 17 | 42 | 10 | 21 | 3 | 22 | 5 | 17 | 3 | 13 | 4 | 12 | 3 | 14 | 4 | 368

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (Day 29)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product.
Time Frame: Up to 28 days post-dose 1 (Day 29)
Population: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants | 96 | 17 | 68 | 17 | 37 | 6 | 25 | 7 | 25 | 3 | 28 | 4 | 31 | 5 | 23 | 4 | 19 | 4

2. Primary Outcome: Number of Participants With Adverse Events (AEs) (28-Day Interval)
Description: as for outcome 1
Time Frame: Up to 28 days post-dose 2 (Day 57 for Cohorts 1, 2a, 2b and 3 [28-Day Interval])
Population: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval
Number analyzed (Participants) | 219 | 39 | 58 | 12 | 55 | 10 | 54 | 12
Participants | 74 | 15 | 22 | 4 | 18 | 4 | 20 | 7

3. Primary Outcome: Number of Participants With Adverse Events (56-day Interval)
Description: as for outcome 1
Time Frame: Up 28 days post-dose 2 (Day 85 for Cohorts 1, 2a, 2b and 3 [56-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 200 | 39 | 59 | 12 | 54 | 10 | 54 | 11
Participants | 58 | 13 | 22 | 4 | 26 | 4 | 22 | 8

4. Primary Outcome: Number of Participants With Adverse Events (84-day Interval)
Description: as for outcome 1
Time Frame: Up to 28 days post-dose 2 (Day 113 for Cohort 1 [84-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval
Number analyzed (Participants) | 98 | 21
Participants | 34 | 7

5. Primary Outcome: Number of Participants With Adverse Events Post-dose 3 (Day 393)
Description: as for outcome 1
Time Frame: Up 28 days post-dose 3 (Day 393)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 34 | 8 | 39 | 9
Participants | 9 | 3 | 14 | 0

6. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 3 years and 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants | 7 | 1 | 7 | 0 | 6 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Immediate Reportable Events (IREs)
Description: The following neuroinflammatory disorders were considered immediate reportable events which had to be reported to the sponsor within 24 hours of becoming aware of the event. Neuroinflammatory disorders included: cranial nerve disorders including paralyses/paresis (example: bell's palsy), optic neuritis, multiple sclerosis, transverse myelitis, guillain-barre syndrome including miller fisher syndrome, bickerstaff's encephalitis and other variants, acute disseminated encephalomyelitis, including site-specific variants (example: non-infectious encephalitis, encephalomyelitis, myelitis, myeloradiculomyelitis), myasthenia gravis and lambert-eaton myasthenic syndrome, immune-mediated peripheral neuropathies and plexopathies, including chronic inflammatory, demyelinating polyneuropathy, multifocal motor neuropathy, and polyneuropathies associated with monoclonal gammopathy, narcolepsy, isolated paresthesia of more than 7 days duration.
Time Frame: Up to 3 years and 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Solicited Local Adverse Events (Day 8)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their diary for 7 days post vaccination. Solicited local AEs were: injection site pain/tenderness, erythema, induration/swelling, itching at the vaccination site.
Time Frame: 7 days post-dose 1 (Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants | 123 | 16 | 121 | 20 | 63 | 11 | 34 | 4 | 35 | 2 | 26 | 3 | 30 | 5 | 26 | 6 | 29 | 5

9. Primary Outcome: Number of Participants With Solicited Local Adverse Events (28-day Interval)
Description: as for outcome 8
Time Frame: Up to 7 days post-dose 2 (Day 36 for Cohort 1, 2a, 2b and 3 [28-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval
Number analyzed (Participants) | 219 | 39 | 58 | 12 | 55 | 10 | 54 | 12
Participants | 126 | 9 | 26 | 2 | 29 | 3 | 22 | 2

10. Primary Outcome: Number of Participants With Solicited Local Adverse Events Post-dose 2 (56-day Interval)
Description: as for outcome 8
Time Frame: Up to 7 days post-dose 2 (Day 64 for Cohort 1, 2a, 2b and 3 [56-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 200 | 39 | 59 | 12 | 54 | 10 | 54 | 11
Participants | 113 | 16 | 25 | 2 | 20 | 3 | 22 | 2

11. Primary Outcome: Number of Participants With Solicited Local Adverse Events (84-day Interval)
Description: as for outcome 8
Time Frame: Up to 7 days post-dose 2 (Day 92 for Cohort 1 [84-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval
Number analyzed (Participants) | 98 | 21
Participants | 57 | 9

12. Primary Outcome: Number of Participants With Solicited Local Adverse Events (Day 372)
Description: as for outcome 8
Time Frame: Up 7 days post-dose 3 (Day 372)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 34 | 8 | 39 | 9
Participants | 18 | 1 | 16 | 3

13. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (Day 8)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. Participants were instructed on how to note signs and symptoms in the diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic events included fever, headache, fatigue/malaise, myalgia, nausea/vomiting, arthralgia and chills.
Time Frame: Up to 7 days post-dose 1 (Day 8)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
Participants | 146 | 27 | 140 | 26 | 75 | 14 | 44 | 7 | 36 | 2 | 29 | 4 | 30 | 5 | 24 | 2 | 23 | 2

14. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (28-Day Interval)
Description: as for outcome 13
Time Frame: Up to 7 days post-dose 2 (Day 36 for Cohorts 1, 2a, 2b and 3 [28-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval
Number analyzed (Participants) | 219 | 39 | 58 | 12 | 55 | 10 | 54 | 12
Participants | 121 | 14 | 32 | 4 | 27 | 3 | 10 | 3

15. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (56-Day Interval)
Description: as for outcome 13
Time Frame: Up 7 days post-dose 2 (Day 64 for Cohort 1, 2a, 2b and 3 [56-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 200 | 39 | 59 | 12 | 54 | 10 | 54 | 11
Participants | 121 | 21 | 26 | 6 | 25 | 6 | 10 | 4

16. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (84-Day Interval)
Description: as for outcome 13
Time Frame: Up 7 days post-dose 2 (Day 92 for Cohort 1 [84-Day Interval])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval
Number analyzed (Participants) | 98 | 21
Participants | 64 | 14

17. Primary Outcome: Number of Participants With Solicited Systemic Adverse Events (Day 372)
Description: as for outcome 13
Time Frame: Up to 7 days post-dose 3 (Day 372)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 34 | 8 | 39 | 9
Participants | 17 | 2 | 18 | 4

18. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Binding Antibody Levels Against Ebola Virus Glycoprotein (EBOV GP) Measured Using Filovirus Animal Non-Clinical Group (FANG) Enzyme-linked Immunosorbent Assay
Description: GMCs of antibodies binding to EBOV GP using FANG ELISA were reported and were measured in ELISA unit per milliliter (EU/mL). Serum samples were collected for analysis of binding antibodies against EBOV GP using FANG ELISA to determine humoral responses following vaccination. For ELISA binding antibody responses, values below the lower limit of quantification (LLOQ) (36.11 ELISA units/mL).
Time Frame: 21-days post-dose 2 (Day 50 for Cohorts 1, 2a, 2b, 3 [28-day interval] , Day 78 for Cohort 1, 2a, 2b, 3 [56-day interval] and Day 106 Cohort 1 [84-day interval]
Population: The per protocol analysis set included all randomized and vaccinated participants, who received both the prime and boost vaccinations (administered not more than 10 days outside the visit window), have immunogenicity data, from baseline and at least one post-vaccination evaluable immunogenicity sample, and have no major protocol violations influencing the immune response.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 225 | 43 | 224 | 44 | 110 | 22 | 59 | 12 | 59 | 12 | 55 | 11 | 55 | 10 | 54 | 12 | 54 | 12
ELISA units/mL
  Day 50 (21 days post-dose 2): number analyzed (Participants) | 171 | 30 | 0 | 0 | 0 | 0 | 58 | 11 | 0 | 0 | 53 | 10 | 0 | 0 | 53 | 12 | 0 | 0
  Day 50 (21 days post-dose 2) | 3085 [2648 to 3594] | NA [NA to NA] — Here, "NA" signifies that the calculated Geometric mean and its 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  |  |  | 4207 [3233 to 5474] | NA [NA to 39] — Here, "NA" signifies that the calculated Geometric mean and its lower limit of 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  | 6993 [5256 to 9303] | NA [NA to 74] — Here, "NA" signifies that the calculated Geometric mean and its lower limit of 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  | 8007 [6321 to 10142] | NA [NA to 82] — Here, "NA" signifies that the calculated Geometric mean and its lower limit of 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |
  Day 78 (21 days post-dose 2): number analyzed (Participants) | 0 | 0 | 136 | 24 | 0 | 0 | 0 | 0 | 59 | 12 | 0 | 0 | 53 | 10 | 0 | 0 | 53 | 11
  Day 78 (21 days post-dose 2) |  |  | 7518 [6468 to 8740] | NA [NA to 53] — Here, "NA" signifies that the calculated Geometric mean and its lower limit of 95% CI were less than LLOQ 36.11 ELISA units/mL) |  |  |  |  | 5283 [4094 to 6817] | NA [NA to NA] — Here, "NA" signifies that the calculated Geometric mean and its 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  | 13532 [10732 to 17061] | 37 [NA to 89] — Here, "NA" signifies that the calculated Geometric mean and its lower limit of 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  | 17388 [12973 to 23306] | NA [NA to NA] — Here, "NA" signifies that the calculated Geometric mean and its 95% CI were less than LLOQ 36.11 ELISA units/mL).
  Day 106 (21 days post-dose 2): number analyzed (Participants) | 0 | 0 | 0 | 0 | 27 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 106 (21 days post-dose 2) |  |  |  |  | 7300 [5116 to 10417] | NA [NA to NA] — Here, "NA" signifies that the calculated Geometric mean and its 95% CI were less than LLOQ 36.11 ELISA units/mL). |  |  |  |  |  |  |  |  |  |  |  |

19. Secondary Outcome: Number of Participants With Serious Adverse Events Post-dose 3
Description: as for outcome 6
Time Frame: Up 28 days post-dose 3 (Day 393)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval
Number analyzed (Participants) | 34 | 8 | 39 | 9
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years and 3 months
Description: Full analysis set included all participants who were randomized and received at least 1 dose of study vaccine (Ad26.ZEBOV, MVA-BN-Filo or placebo).
Arm/Group | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval | Cohort 1: Placebo, Placebo, 84-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2a: Placebo, Placebo, 28-Day Interval | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2a: Placebo, Placebo, 56-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 2b: Placebo, Placebo, 28-Day Interval | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 2b: Placebo, Placebo, 56-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval | Cohort 3: Placebo, Placebo, 28-Day Interval | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval | Cohort 3: Placebo, Placebo, 56-Day Interval
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/43 | 0/224 | 0/44 | 0/110 | 0/22 | 1/59 | 0/12 | 0/59 | 0/12 | 1/55 | 0/11 | 0/55 | 0/10 | 0/54 | 0/12 | 0/54 | 0/12
Serious Adverse Events (participants affected / at risk) | 7/225 | 1/43 | 7/224 | 0/44 | 6/110 | 0/22 | 1/59 | 0/12 | 1/59 | 0/12 | 1/55 | 0/11 | 0/55 | 0/10 | 1/54 | 0/12 | 0/54 | 1/12
Other Adverse Events (participants affected / at risk) | 94/225 | 17/43 | 80/224 | 21/44 | 43/110 | 12/22 | 24/59 | 9/12 | 28/59 | 5/12 | 29/55 | 5/11 | 33/55 | 6/10 | 27/54 | 9/12 | 22/54 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval (N=225) | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval (N=43) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval (N=224) | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval (N=44) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval (N=110) | Cohort 1: Placebo, Placebo, 84-Day Interval (N=22) | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=59) | Cohort 2a: Placebo, Placebo, 28-Day Interval (N=12) | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=59) | Cohort 2a: Placebo, Placebo, 56-Day Interval (N=12) | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=55) | Cohort 2b: Placebo, Placebo, 28-Day Interval (N=11) | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=55) | Cohort 2b: Placebo, Placebo, 56-Day Interval (N=10) | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=54) | Cohort 3: Placebo, Placebo, 28-Day Interval (N=12) | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=54) | Cohort 3: Placebo, Placebo, 56-Day Interval (N=12)
Dolichocolon (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniere's Disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anembryonic Gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 28-Day Interval (N=225) | Cohort 1: Placebo, Placebo, Placebo, 28-Day Interval (N=43) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, Ad26.ZEBOV, 56-Day Interval (N=224) | Cohort 1: Placebo, Placebo, Placebo, 56-Day Interval (N=44) | Cohort 1: Ad26.ZEBOV, MVA-BN-Filo, 84-Day Interval (N=110) | Cohort 1: Placebo, Placebo, 84-Day Interval (N=22) | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=59) | Cohort 2a: Placebo, Placebo, 28-Day Interval (N=12) | Cohort 2a: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=59) | Cohort 2a: Placebo, Placebo, 56-Day Interval (N=12) | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=55) | Cohort 2b: Placebo, Placebo, 28-Day Interval (N=11) | Cohort 2b: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=55) | Cohort 2b: Placebo, Placebo, 56-Day Interval (N=10) | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 28-Day Interval (N=54) | Cohort 3: Placebo, Placebo, 28-Day Interval (N=12) | Cohort 3: Ad26.ZEBOV, MVA-BN-Filo, 56-Day Interval (N=54) | Cohort 3: Placebo, Placebo, 56-Day Interval (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 14 | 1 | 8 | 4 | 2 | 2 | 2 | 2 | 6 | 1 | 2 | 0 | 3 | 1 | 1 | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Infection Parasitic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0
Malaria (Infections and infestations) | 16 | 2 | 12 | 5 | 6 | 2 | 1 | 0 | 3 | 0 | 3 | 1 | 8 | 1 | 7 | 2 | 4 | 0
Nasopharyngitis (Infections and infestations) | 8 | 4 | 11 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 4 | 2 | 1 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 7 | 0 | 2 | 1 | 4 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 1 | 18 | 3 | 9 | 3 | 7 | 1 | 3 | 1 | 6 | 0 | 3 | 2 | 0 | 1 | 4 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Blood Potassium Decreased (Investigations) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Sodium Decreased (Investigations) | 9 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Blood Urea Decreased (Investigations) | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Monocyte Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases Increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 6 | 1 | 7 | 0 | 4 | 1 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 3 | 3 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 5 | 0 | 2 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 15 | 4 | 8 | 3 | 7 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 3 | 1 | 1 | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 2 | 3 | 2 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A total of 259 participants in Cohort 1 either did not receive dose 2 (N=52) or received dose 2 outside of their protocol-defined interval (N=207), mainly due to the study pause resulting in a reduced precision for the immunogenicity estimates in the Per Protocol Analysis Set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT02564523/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT02564523/SAP_001.pdf